CLINICAL TRIAL: NCT01824485
Title: Best Effect of Viscosupplementation With Hyaluronic Acid and Triamcinolone in Patients With Knee Osteoarthritis. Prospective Randomized Study Between Two Different Applications Regimens
Brief Title: Comparison of Two Application Regimens for Viscosupplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPPesq 0199/11
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee; Viscosupplementation; Clinical Trial
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Experimental): Patients from Group 2 will receive an intra-articular injection of 1 ampoule (2ml) of OSTEONIL®, on a weekly basis, for 3 weeks (total of 3 injections)
  Interventions: Drug: viscosupplementation 1+1+1
- Group 1 (Experimental): Patients from Group 1 will receive a single intra-articular injection of 3 ampoule (6ml) of OSTEONIL®
  Interventions: Drug: viscosupplementation 3 at once

INTERVENTIONS:
Drug: viscosupplementation 1+1+1 — intra-articular injection with 1 ampoule per week for 3 weeks
  Other Names: 1+1+1
  Arms: Group 2
Drug: viscosupplementation 3 at once — single intra-articular injection with 3 ampoules
  Arms: Group 1

SUMMARY:
Viscosupplementation by intra-articular injection of hyaluronate products has recently gained popularity as a treatment modality of gonarthritis.There is not, however, a consensus on the best method.Our objective is to evaluate what is the best dosage of viscosupplementation with hyaluronic acid (OSTEONIL®) associated with 1 ml (20 mg) of triamcinolone hexacetonide. One hundred and four patients with knee osteoarthritis (KOA) were divides into 2 groups of 52 patients each to receive either a single application of 3 ampoules of OSTEONIL® + 1ml of Hexacetonide of triamcinolone or three applications of 1 ampoule of OSTEONIL®, one per week for three weeks + 1ml of Hexacetonide of triamcinolone only in the first injection. Primary endpoint was clinical results expressed by Visual Analogic Scale of pain (VAS), Western Ontario and Mcmaster Universities (WOMAC) and Lequesne questionaires at one, three, six and 12 months after the procedure

DETAILED DESCRIPTION:
Viscosupplementation by intra-articular injection of hyaluronate products has recently gained popularity as a treatment modality of gonarthritis. Hyaluronic Acid is responsible for the elasticity and viscosity of the synovial fluid, protecting the joint. Biopsy studies show that besides the gain in pain and function, viscosupplementation may lead to structural changes of the cartilage. Currently there are several studies on the effect of intra-articular injection of hyaluronic acid in gonarthritis. There is not, however, a consensus on the best method. Regarding the substance to be injected, corticosteroids alone exhibit rapid results, but poor durability. Viscosupplementation shows more consistent results. However, especially when using derivatives with higher molecular weight hyaluronan, there is a significant number of patients that present an acute synovial reaction to viscosupplementation specially in the first cycle of three injections. The association triamcinolone injection with hyaluronic acid decreases the complaints in the first month of treatment. Our objective is to evaluate what is the best dosage of viscosupplementation with hyaluronic acid (OSTEONIL®) associated with 1 ml (20 mg) of triamcinolone hexacetonide by comparing two groups of patients with knee OA, the first with a single application of 3 ampoules and second with three applications, one per week for three weeks. One hundred and four knee osteoarthritis (KOA) patients, which are currently in usual care for KOA at the Osteometabolic Group - Department of Orthopedics and Traumatology - University of São Paulo General Hospital - will be assessed. After signing the informed consent, participants will respond WOMAC™, Lequesne™, VAS, SF-36 (quality of life) and subjective IKDC (International Knee Documentation Committee). The questionnaires and functional assessment will be performed before the procedure infiltration with 1month, 3 months, 6 months and 1 year of intervention.Twenty Patients will be submitted to evaluation using force platform and balance NeuroCom ®, with the following tests: weight support during the squat (weight bearing squat (WBS), one-leg support (unilateral stance (U.S.), from sitting to foot (sit to stand - STS). Previously, at 1 month, 3 month, 6 month and 12 months after the intervention.

Frontal weight-bearing, profile and axial radiographs will be performed to radiologically assess participants' knees.Patients will be randomly divided into two groups of 54 patients, (groups 1 and 2). Patients in group 1 (G1) will be submitted to viscosupplementation with 1 application of 3 vials of hyaluronic acid 20mg/2ml (OSTEONIL®) and 1 ml (20 mg) triamcinolone, whereas group 2 patients will be submitted to viscosupplementation with three applications of one ampoule of hyaluronic acid 20 mg/2ml (one per week for three weeks), with the first application of OSTEONIL® with 1 ml (20 mg) triamcinolone.

ELIGIBILITY:
Inclusion Criteria:

* Met the American College of Rheumatology criteria for hip osteoarthritis
* No knee intraarticular injections in the last 6 months

Exclusion Criteria:

* Severe reaction to the procedure

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
WOMAC | 6 months
  Pain and function assessment with WOMAC questionaire
VAS | 6 months
  Pain assessment with Visual Analogic Scale (VAS)
LEQUESNE | 6 months
  Pain and function assessment with Lequesne questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, Phd, Principal Investigator — FMUSP
Locations (1):
- Instituto de Ortopedia e Traumatologia HC-FMUSP, São Paulo, São Paulo, Brazil